CLINICAL TRIAL: NCT04853251
Title: A Phase IV, Multicenter, Open-label Study to Assess Corneal Endothelial Cells in Patients With Neovascular Age-related Macular Degeneration Treated With the Port Delivery System With Ranibizumab (PDS)
Brief Title: A Study Assessing Corneal Endothelial Cells in Participants With Neovascular Age-related Macular Degeneration (nAMD) Treated With the Port Delivery System With Ranibizumab (PDS)
Acronym: Belvedere
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML43000
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Masking Description: The BVCA examiner will be masked as best as possible to participant study eye assignment and study visit type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- SUSVIMO (Experimental): Participants will have the PDS implant (filled prior to implantation with approximately 20 microlitres [uL] of the 100 milligrams/millilitres [mg/ml] formulation of ranibizumab [approximately 2 milligrams (mg) dose of ranibizumab]) surgically inserted in the study eye at the Day 1 visit following their enrollment visit. After the initial fill of the implant with ranibizumab, participants will receive implant refill-exchanges at fixed Q24W intervals.
  Interventions: Device: PDS Implant With Ranibizumab 100 mg/ml; Drug: LUCENTIS (Ranibizumab Injection)

INTERVENTIONS:
Device: PDS Implant With Ranibizumab 100 mg/ml — Ranibizumab 100 mg/mL will be delivered via PDS
Drug: LUCENTIS (Ranibizumab Injection) — Ranibizumab (0.5 mg intravitreal [IVT] injections of 10 mg/mL formulation) will be used in the study eye as supplemental treatment. If a participant discontinues study treatment, he/she may start receiving IVT ranibizumab injections in the study eye, per investigator's discretion.

SUMMARY:
This study will assess corneal endothelial cells in participants with nAMD treated with PDS refilled every 24 weeks (Q24W).

ELIGIBILITY:
Inclusion Criteria

Ocular Inclusion Criteria:

* Diagnosis of nAMD prior to screening as determined by the investigator
* Difference of <10% in ECD at screening between the 2 eyes as measured by specular microscopy and determined by the independent reading center
* Availability of historical visual acuity (VA) data and spectral-domain optical coherence tomography (SD-OCT). Additionally, fluorescein angiography or color fundus photography can both be used to support participant eligibility per protocol at investigator discretion
* Availability of comprehensive historical anti-vascular endothelial growth factor (VEGF) injection data, including agent administered and date of administration from the time of diagnosis, or for at least 2 years prior to screening if diagnosis was made more than 2 years before screening
* Response to at least two prior anti-VEGF IVT injections as determined by the investigator based on the following:

  * Overall decrease in nAMD disease activity detected on historical or screening OCT
  * Stable or improved best-corrected visual acuity (BCVA)
* BCVA of 34 letters (approximate 20/200 Snellen equivalent) or better, using Early Treatment of Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters at screening and enrollment
* All subtypes of nAMD lesions are permissible
* nAMD lesions at the time of diagnosis must involve the macula
* Sufficiently clear ocular media and adequate pupillary dilation to allow for clinical examination and analysis and grading by the central reading center of SD-OCT images

Exclusion Criteria

Prior Ocular Treatment

Study Eye:

* Prior treatment with external-beam radiation therapy or transpupillary thermotherapy
* Previous treatment with verteporfin injection (PDT) or corticosteroid IVT injection within 2 years of screening
* Previous laser (except PDT as stated above) used for age related macular degeneration (AMD) treatment
* History of corneal transplant
* History of conjunctival surgery in the superotemporal quadrant
* History of intraocular inflammation following anti-VEGF injection

Either Eye:

* Previous PDS implantation
* Previous intraocular surgery (including cataract surgery) within 6 months of study enrollment
* Prior vitrectomy surgery, submacular surgery, or other surgical intervention for age-related macular degeneration (AMD)
* Prior pars plana vitrectomy surgery
* Previous intraocular device implantation, excluding intraocular lenses
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery
* Prior participation in a clinical trial involving any intravitreal agents that are not approved at time of screening
* Intraocular laser therapy, including selective laser trabeculoplasty, yttrium-aluminum garnet (YAG), prophylactic peripheral iridotomy within 1 year of screening, or YAG capsulotomy within 3 months of screening
* Contact lens wear in either eye within 2 months of screening
* Any prior penetrating ocular trauma
* Any prior ocular blunt trauma affecting corneal or retinal health in the opinion of the investigator, or any ocular blunt trauma within 6 months of screening
* History of corneal transplantation, including partial-thickness corneal grafts
* Prior treatment with brolucizumab
* Prior treatment with external-beam radiation therapy or brachytherapy
* History of hypersensitivity to ranibizumab or any excipients of Susvimo

Macular Neovascularization Lesion (MNV) Characteristics

Study Eye:

* Subretinal hemorrhage that involves the center of the fovea, if the hemorrhage is greater than 0.5-disc area [1.27 square millimeters (mm^2)] in size
* Subfoveal fibrosis or subfoveal atrophy

Either Eye:

* MNV due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* MNV masquerading lesions (e.g., cone dystrophy, adult vitelliform dystrophy, pattern dystrophy)

Current or Historical Ocular Conditions

Study Eye:

* Retinal pigment epithelial tear
* Retinal tears or peripheral retinal breaks on depressed fundus exam that are untreated, or treated within the 3 months prior to study enrollment
* Current vitreous hemorrhage
* Current or history of retinal detachment
* Previous violation of the posterior capsule is also an exclusion criterion unless it occurred as a result of YAG laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
* Spherical equivalent of the refractive error demonstrating more than 8 diopters of myopia or evidence of pathologic myopia on depressed fundus examination
* Preoperative refractive error that exceeds 8 diopters of myopia, for participants who have undergone prior refractive or cataract surgery
* Spherical equivalent of the refractive error demonstrating more than 5 diopters of hyperopia
* Preoperative refractive error that exceeds 5 diopters of hyperopia, for participants who have undergone prior refractive or cataract surgery
* Uncontrolled ocular hypertension or glaucoma and any such condition the investigator determines may require a glaucoma-filtering surgery during a patient's participation in the study
* Scleral pathology in the superotemporal quadrant (e.g., scleral thinning or calcification)
* Conjunctival pathologies in the superotemporal quadrant
* History or presence of severe posterior blepharitis, recurrent chalazia or hordeolum, severe dry eye syndrome, or severe allergic conjunctivitis
* Ectropion, entropion or other impairment of the upper or lower eyelid impacting lid functionality needed to protect the ocular surface from exposure
* Trichiasis
* Corneal neuropathy
* Lagophthalmos or incomplete blink
* Active or history of facial nerve palsy/paresis

Fellow (Non-Study) Eye:

• Concurrent or history of PDS implantation

Either Eye:

* Aphakia or absence of the posterior capsule
* Any concurrent intraocular condition that would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results
* Corneal ECD ≤1500 cells/mm2 in either eye at screening as determined by the independent reading center
* Fuchs endothelial corneal dystrophy Grade ≥ 2
* Previous corneal endothelial cell damage, including from blunt or surgical trauma
* Any ocular condition that precludes obtaining an analyzable specular microscopy image
* Active or history of corneal edema
* Active or history of corneal dystrophies
* Active or history of iridocorneal endothelial syndrome
* Active or history of pseudoexfoliation syndrome
* Active or history of herpetic keratitis or kerato-uveitis
* Any active or history of uveitis
* Active intraocular inflammation
* Active or history of keratitis, scleritis, or endophthalmitis
* Active ocular or periocular infection
* Active or history of Sjogren's syndrome or keratoconjunctivitis sicca
* Active or history of floppy eyelid syndrome
* Active or history of chronic eye rubbing
* Active thyroid eye disease

Concurrent Systemic Conditions:

* History of uncontrolled blood pressure
* Active or history of autoimmune diseases such as rheumatoid arthritis, lupus, granulomatosis with polyangiitis (Wegener's)
* History of stroke within the last 3 months prior to screening
* Uncontrolled atrial fibrillation within 3 months of screening
* History of myocardial infarction within the last 3 months prior to screening
* History of other disease, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab or placement of the implant and that might affect interpretation of the results of the study or renders the patient at high risk of treatment complications, in the opinion of the investigator
* Current active systemic infection
* Use of any systemic anti-VEGF agents
* Chronic use of oral corticosteroids
* Active cancer within 12 months of enrollment except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of ≤ 6 and a stable prostate-specific antigen for > 12 months
* Previous participation in any non-ocular (systemic) disease studies of investigational drugs within 1 month prior to screening (excluding vitamins and minerals)
* Use of antimitotic or antimetabolite therapy within 30 days or 5 elimination half-lives of the screening visit
* Requirement for continuous use of any medications or treatments indicated as prohibited therapy
* Pregnant or breastfeeding, or intention to become pregnant during the study
* Women of childbearing potential must have a negative urine pregnancy test result within 28 days prior to initiation of study treatment. If the urine pregnancy test is positive, it must be confirmed by a serum pregnancy test

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Corneal Endothelial Cell Density (ECD) From Baseline at Week 48 in the Study Eye as Compared With the Fellow Eye, as Assessed by Specular Microscopy | Baseline, Week 48

SECONDARY OUTCOMES:
Percent Change in Corneal ECD From Baseline at Week 24 in the Study Eye as Compared With the Fellow Eye | Baseline, Week 24
Percent Change in the Coefficient of Variation (CV) of Corneal Endothelial Cell Area From Baseline at Weeks 24 and 48 in the Study Eye as Compared With the Fellow Eye | Baseline, Week 24, Week 48
Percent Change in Hexagonal Cells (HEX) From Baseline at Weeks 24 and 48 in the Study Eye as Compared With the Fellow Eye | Baseline, Week 24, Week 48
Percentage of Participants With Ocular Serious Adverse Events (SAEs) and Severity of SAEs | Day 1 up to approximately Week 52
Percentage of Participants With Ocular Adverse Events of Special Interests (AESIs) and Severity of Ocular AESIs | Day 1 to Week 52
Duration of Ocular AESIs | Day 1 to Week 52
Percentage of Participants With Ocular AESIs During the Postoperative Period | Baseline up to 37 days of initial implantation
Percentage of Participants With Ocular AESIs During the Intermediate Postoperative Period | 38 to 93 days after implantation
Percentage of Participants With Ocular AESIs During the Follow-up Period | Week 52
  The investigator will follow each adverse event (AE) until the event has resolved to baseline grade or better, the event is assessed as stable by the investigator, the participant is lost to follow-up, or the participant withdraws consent.
Percentage of Participants With Adverse Device Effects (ADEs) | Day 1 to Week 52
Number of Participants with Anticipated Serious Adverse Device Effects (ASADEs) and Severity of ASADEs | Day 1 to Week 52
Duration of ASADEs | Day 1 to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (50):
- United States (50):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina Associates of Southern California, Huntington Beach, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retinal Consultants Med Group, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - Macula Retina Vitreous Research Institute, Torrance, California
  - Southwest Retina Consultants, Durango, Colorado
  - Advanced Vision Research Institute, Longmont, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Retina Specialty Institute, Pensacola, Florida
  - Ft Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Wilmer Eye Institute Johns Hopkins University, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - VitreoRetinal Surgery, PLLC., Minneapolis, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Seeta Eye Centers, Poughkeepsie, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - Fargo Retina Consultants, Fargo, North Dakota
  - Cincinnati Eye Institute, Blue Ash, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Erie Retina Research, Erie, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Palmetto Retina Center, Florence, South Carolina
  - Palmetto Retina Center, LLC, West Columbia, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Panhandle Eye Group LLP Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Schertz, Texas
  - Retina Associates of Utah, PLLC, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing